CLINICAL TRIAL: NCT02113735
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Safety and Efficacy Study of H.P. Acthar® Gel (Acthar) in Subjects With Acute Respiratory Distress Syndrome (ARDS)
Brief Title: Safety and Efficacy Study of Acthar in Subjects With ARDS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: A company decision was made not to proceed with the study.
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QSC01-ARDS-01
Record Dates: First submitted 2014-04-08; First posted 2014-04-15 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: ARDS; Acute Respiratory Distress Syndrome; Acthar; ACTH; H.P. Acthar Gel
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Experimental): H.P. Acthar® Gel , 64 U, 0.8 mL daily
  Interventions: Drug: H.P. Acthar® Gel (repository corticotropin injection)
- Group 2 (Placebo Comparator): Placebo, 0.8 mL, daily
  Interventions: Drug: Placebo
- Group 3 (Experimental): H.P. Acthar® Gel , 32 U, 0.4 mL, 2x daily
  Interventions: Drug: H.P. Acthar® Gel (repository corticotropin injection)
- Group 4 (Placebo Comparator): Placebo, 0.4 mL, 2x daily
  Interventions: Drug: Placebo
- Group 5 (Experimental): H.P. Acthar® Gel , 16 U, 0.2 mL, 2x daily
  Interventions: Drug: H.P. Acthar® Gel (repository corticotropin injection)
- Group 6 (Placebo Comparator): Placebo, 0.2 mL, 2x daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: H.P. Acthar® Gel (repository corticotropin injection)
  Other Names: Acthar
  Arms: Group 1; Group 3; Group 5
Drug: Placebo
  Arms: Group 2; Group 4; Group 6

SUMMARY:
This study is being performed to evaluate the potential efficacy and safety of Acthar as a treatment for moderate-severe Acute Respiratory Distress Syndrome (ARDS). Approximately 210 subjects will be randomized to 1 of 6 possible treatment groups in a 3:2:3:2:3:2 ratio. Study medication (SM) will be administered via subcutaneous (SC) injection for 4 weeks using a blinded gradually tapering regimen, and subjects will be followed for 60 days post-randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥ 18 years.
2. ARDS as defined by:

   * PaO2 /FiO2 ≤ 200 mmHg with PEEP ≥ 5cm H2O.
   * Bilateral opacities on chest radiography not explained by atelectasis, effusions, nodules, or preexisting disease.
   * Requirement for positive pressure ventilation via an endotracheal tube.
   * Respiratory failure not fully explained by cardiac failure or fluid overload. If no identifiable risk factor for ARDS is identified, left atrial hypertension must be excluded by objective measures (e.g. transthoracic echocardiogram).
   * Criteria 2a, 2b, and 2c must occur within the same 24 hr period.
3. Enrollment between 24 hours and 10 days after ARDS criteria are met.

Exclusion Criteria:

1. Subject unwilling to receive or intolerant of SC injections.
2. Subject, surrogate, or physician not committed to full supportive care. A "Do Not Resuscitate" (DNR) order alone without other limitations of care does not require study exclusion.
3. Moribund subject with death perceived to be imminent. For the purposes of this study, moribund is defined by a requirement for ≥ 2 high dose vasopressors AND acute organ failures in ≥ 3 organs for ≥ 24 hours prior to study entry.
4. Home mechanical ventilation (noninvasive ventilation or via tracheotomy) except for continuous positive airway pressure or bi-level positive airway pressure (CPAP/BIPAP) used solely for sleep-disordered breathing prior to onset of ARDS.
5. Known contraindication to Acthar per package insert Section 4 (Appendix C): scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of peptic ulcer, congestive heart failure, uncontrolled hypertension, primary adrenocortical insufficiency, or adrenal cortical hyperfunction.
6. Gastrointestinal/Hepatic: History of chronic active hepatitis, active Hepatitis B or acute or chronic Hepatitis C infection, OR moderate-severe chronic liver disease as defined by a Child-Pugh Score > 11(http://gihep.com/calculators/hepatology/child-pugh-score/), OR any evidence of hemodynamically significant active gastrointestinal (GI) bleeding.
7. Any subject with signs or symptoms concerning for an active infection that has not been treated for > 48 hours prior to randomization with either empiric broad-spectrum or pathogen-directed anti-microbial therapy.
8. Immune System: Known immune-compromised status, including but not limited to individuals who have undergone organ transplantation or who are known to be positive for the human immunodeficiency virus (HIV).
9. Burns >20% total body surface area, or any burn injury accompanied by smoke inhalational injury.
10. Major surgery within 48 hours before randomization, OR evidence of currently active bleeding postoperatively, OR plan for any major surgery during the study period.
11. Administration of any other investigational drug or participation in an interventional clinical research study for ARDS within 30 days of planned randomization or during the 60 day study duration.
12. Presence of any other clinically significant disease or disorder (including those listed in Appendix C package insert Section 5 [Warnings and Precautions]) which, in the opinion of the Investigator (by its nature or by being inadequately controlled), might put the subject at risk due to participation in the study, or may influence the results of the study or the subject's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08 (Estimated); Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Number of ventilator-free days (subjects alive and breathing without assistance for ≥ 48 hr) by Day 28 after randomization | 60 days (28 days of treatment with a 32 day follow-up period)

SECONDARY OUTCOMES:
Mortality at Day 28 and Day 60 | 60 days (28 days of treatment with a 32 day follow-up period)
Number of ICU-free and hospital free days for all subjects who survive to ICU and hospital discharge, respectively | 60 days (28 days of treatment with a 32 day follow-up period)
Number of extra-pulmonary organ failure-free days | 60 days (28 days of treatment with a 32 day follow-up period)
Change in PaO2/FiO2 ratio and oxygenation index (OI) from baseline for subjects on mechanical ventilation | 60 days (28 days of treatment with a 32 day follow-up period)
Change in Systemic Organ Failure Assessment Score (SOFA) score from baseline. | 60 days (28 days of treatment with a 32 day follow-up period)
Number of treatment-emergent serious adverse events | 60 days (28 days of treatment with a 32 day follow-up period)
Number, severity and site of new infections developing at least 48 hr after initiation of Study Medication | 60 days (28 days of treatment with a 32 day follow-up period)
Proportion of subjects who discontinue treatment because of serious safety concerns | 60 days (28 days of treatment with a 32 day follow-up period)